CLINICAL TRIAL: NCT06901063
Title: Research of the Sonographic Anatomy of Interscalene Brachial Plexus
Brief Title: Research of Brachial Plexus Anatomy
Acronym: Soana-ibp
Status: Completed | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Xiaoyu Yang, MD, Huashan Hospital
Other Study IDs: 2025-yxy-1
Record Dates: First submitted 2025-03-23; First posted 2025-03-28 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Brachial Plexus Injury; Ultrasound
Keywords: Brachial plexus; Nerve block; Ultrasound
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The study group: The recruited patients will be included in this group
  Interventions: Device: ultrasound

INTERVENTIONS:
Device: ultrasound — Using ultrasound probe to scan and record the bilateral interscalene brachial plexus

SUMMARY:
The research aims at analyzing the sonographic anatomy characteristics of the interscalene brachial plexus.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status class I or II
* Scheduled for elective surgery

Exclusion Criteria:

* Skin lesion or infection of neck
* Any known peripheral neuropathy
* Brachial nerve plexus injury
* Previous injury or operation on neck
* Pregnancy or breast feeding
* Allergic to ultrasound gel

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospectively collect ultrasound video of interscalene brachial plexus from existed departmental database.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
The distribution of the number of visible bundles in C6 nerve root | immediately after the procedure
  The percentage of one, two and multiple nerve bundles which composing the C6 nerve root

SECONDARY OUTCOMES:
The distribution of the number of visible bundles in C5 nerve root | immediately after the procedure
  The percentage of one, two and multiple nerve bundles which composing the C5 nerve root
The distribution of the number of visible bundles in C7 nerve root | immediately after the procedure
  The percentage of one, two and multiple nerve bundles which composing the C7 nerve root

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No